CLINICAL TRIAL: NCT01129154
Title: An Open Label Multicentric Phase II Study of Panitumumab (Vectibix®) in Cutaneous Squamous Cell Carcinoma (SCC)
Brief Title: Panitumumab (Vectibix®) in Cutaneous Squamous Cell Carcinoma (SCC)
Acronym: PASCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Cliniques Universitaires UCL de Mont-Godinne, Dr Joseph Kerger (Unknown); Cliniques Saint-Pierre Ottignies, Dr Lionel Duck (Unknown)
Responsible Party: Baurain Jean-François, Cliniques universitaires Saint-Luc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Luc 09-002
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Squamous cell carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- panitumumab (Experimental): Patients will receive six infusions of panitumumab every 2 weeks for the first cycle.
  Interventions: Drug: infusions of Panitumumab

INTERVENTIONS:
Drug: infusions of Panitumumab — Patients will receive six infusions of Panitumumab 6 mg/kg every 2 weeks or until progression if earlier.
  Other Names: Vectibix®

SUMMARY:
Squamous Cell Carcinoma (SCC) is one of the most common malignancies in caucasian population. The effect of the immune system on the development of skin tumors has been demonstrated in transplant patients taking immunosuppressive agents (65 fold risk increase). It has been reported that activation of EGFR and RAS signaling pathways play an important role in disease progression maybe through downregulation of the immune system.

The investigators want to treat unresectable SCC patients with an antibody against EGFR (Vectibix®, panitumumab). This antibody induces tumor regression in metastatic colorectal cancer and has been approved as single agent for this indication.

The investigators want to measure the response rate but also analyze the modification of expression profile of some key proteins involved or supposed to be involved in the signaling pathways of EGFR and in the regulation of the immune system. Chemokines such as CCL27 have been shown to play a critical role in the skin-associated immune response by regulating T cell homing. Pivarcsi et al have reported that downregulation of CCL27 is mediated by activation of EGFR/RAS/MAPK signaling pathways.

DETAILED DESCRIPTION:
This is an open-label, multicentric study of 17 patients with skin squamous cancer cell.

Eligible patients should not be suitable for immediate surgery. If they have only one tumor, it should be greater than 3 cm2 in order to allow multiple biopsies.

Patients will receive six infusions of Panitumumab 6 mg/kg every 2 weeks or until progression if earlier.

Patients will be assessed at baseline, at week 6 and then every 12 weeks till progression. In addition to clinical examination, evaluation tools will include photography and CT-scan, MRI or PET-scan.

Skin and tumor biopsies will be performed during first cycle at baseline and at days 2, 4, 8, 43, 85. Blood collections for translational research will be done during first cycle at baseline and at days 2, 4, 8,15, 43, 85. Blood collection for hematology and chemistry assessment will be done each 4weeks.

Patients presenting with a stable disease or a tumor response at week 12 will be eligible for maintenance cycles consisting in an infusion of panitumumab every 2 weeks till progression.

ELIGIBILITY:
Inclusion criteria

* Patient with histologically confirmed diagnosis of SCC.
* Patient must not be candidate to direct curative surgery.
* Tumor evaluation by photography with a ruler and CT-scan, MRI or PET-scan must be performed before enrollment.
* Age ≥ 18 years.
* Karnofsky Performance status (KPS) ≥70.
* Normal laboratory values:

  * Platelet count ≥100x103/μL
  * Leucocyte count ≥ 3x103/μL
  * Hemoglobin ≥ 9 g/dL
  * ASAT and ALAT ≤ 2.5xUNL
  * Serum creatinine ≤1.5xUNL
  * Total bilirubin ≤ 1.5xUNL
  * Magnesium ≥ Lower Normal Limit (LLN)
  * Calcium ≥ Lower Normal Limit (LLN)
* Patient should agree to perform biopsies and blood collections for translational research.
* Signed informed consent from the patient or legal representative must be obtained.

Exclusion criteria

* Clinically significant cardiovascular disease (including cardiac insufficiency NYHA grade III and IV, unstable angina, arrythmia, myocardial infarction, symptomatic congestive heart failure)in the past 12 months before enrollment.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* No prior chemotherapy.
* Prior anti-EGFR therapy.
* Radiation within four weeks prior to trial entry.
* Subject pregnant or breastfeeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months after the end of treatment.
* The patient has (or has had) previous or concomitant malignancies at other sites within last 5years, except effectively treated malignancy that is considered by the investigator highly likely to have been cured.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | via imaging every 12 weeks
  To measure the efficacy of Panitumumab for SCC in terms of Overall Response Rate (ORR). Overall Response Rate (ORR) is defined as the sum of complete and partial tumour responses seen, divided by the total number of evaluable patients.

SECONDARY OUTCOMES:
To assess the safety profile of panitumumab in SCC | at each visit
  Proportion of all adverse events will be reported. CTC scale 3.0 will be used with the exception of skin- or nail-related toxicities, which must be graded using CTC version 3.0 with modifications (Appendix E). Patients will be followed for safety until closure of study.
Time to treatment failure (TTF)and Time to treatment progression TTP | via imaging, every 12 weeks
  Time to treatment failure (TTF) is defined as the time from date of first dose of study medication to first occurrence of any following event : documentation of objective tumor progression, toxicities requiring prematurely stop of treatment or death. TTF will be calculated according to the Kaplan-Meier technique. Time to Progression will also be calculated. Subjects without evidence of progression at the end of follow up will be considered as censored.
To measure the duration of response. | via imaging, every 12 weeks
  Duration of overall response will be measured according RECIST guidelines version 1.1 Duration of response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
To explore the gene expression profiles in SCC under panitumumab treatment (i.e CCL27, EGFR,…). | Skin and tumor biopsies will be performed at baseline and at days 2, 4, 8, 43, 85. Blood will be collected at baseline and at days 2, 4, 8, 43, 85
  Results will be presented as proportion of each expression type.

CONTACTS AND LOCATIONS:
Overall Officials: Baurain Jean-Francois, Md,PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (3):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc Université Catholique de Louvain, Brussels, Brussels Capital
  - Cliniques Universitaires UCL, Mont Godinne
  - Cliniques Saint-Pierre, Ottignies